CLINICAL TRIAL: NCT02577445
Title: The remedē® System (Respiratory Rhythm Management™ Device) for the Treatment of Central Sleep Apnea in Daily Practice
Brief Title: The remedē® System for the Treatment of Central Sleep Apnea in Daily Practice
Acronym: TREAT-CSA
Status: Terminated | Type: Observational
Why Stopped: Commercial distribution of the remedē System stopped by LivaNova.
Sponsor: LivaNova (Industry)
Collaborators: Respicardia, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NVNS03
Record Dates: First submitted 2015-09-25; First posted 2015-10-16 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Sleep Apnea; Central Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Central

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CSA patients without remedē system: For all patients diagnosed with CSA who will not move forward with remedē® system therapy, the intention is to obtain information on their alternate therapy, if any, and safety information, including all cause mortality and all cause hospitalizations during phone calls at 6, 12 and 24 months after enrollment.
- CSA patients with remedē system: For all patients diagnosed with CSA and referred for implant / or have already been implanted with remedē system, information from the implant procedure will be collected.
  Patients will be asked to complete quality of life questionnaires at baseline and during follow-up visits.
  Patients will be evaluated at the time of therapy activation which may be followed by one or more titration visits. Patient follow-ups will be programmed at 6 and 12 months, and yearly, up to 5 years post-implant, until the last patients reach their 2-year follow-up.
  Echocardiogram for patients with reduced ejection fraction (≤ 45%) and follow-up respiratory polygraphy are considered standard of care, however, to ensure sufficient data, related to the study objectives, are being collected, baseline and 12-months echocardiogram for a subgroup of patients and respiratory polygraphy at 12-month follow-up for all patients must be done when participating in this study:

SUMMARY:
The aim of this post market study is to assess the impact of sleep-disordered breathing on the well-being of patients according to the treatment chosen, i.e. with or without implantation of the remedē® system to treat sleep-disordered breathing.

DETAILED DESCRIPTION:
The sponsor of this study, LivaNova, has a partnership with Respicardia, Inc who has developed a battery-powered implantable device that treats central sleep apnea. The device is used with a lead that delivers the stimulation therapy which causes the patient to breathe with a regular rhythm and an optional lead that senses breathing. This combination is called the remedē® system.

The aim of this study is

1. to collect data in order to get a better understanding of the characteristics and/or symptoms related to central sleep apnea
2. to collect safety information of all patients diagnosed with central sleep apnea
3. to obtain additional short and lang term information on the safety and performance of the remedē® system, including an evaluation if there's an impact on the quality of life of patients treated with the the remedē® system in daily practice.

The information obtained from this study may provide better insight on the symptoms related to central sleep apnea, risk factors related to central sleep apnea therapy and use of the remedē® system which may help to treat other patients with potential sleep disordered breathing more appropriately.

Approximately 300 patients (to be) implanted with the remedē® system will participate in this study at approximately 40 sites in Europe. For this purpose the investigators aim to screen approximately 1500 patients with sleep-disordered breathing. Also patients diagnosed with central sleep apnea, but not receiving the device will be followed through phone calls for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients screened for sleep disordered breathing
* Age > 18 years
* Signed Ethics Committee approved informed consent

Implant Inclusion criteria

* Diagnosis of moderate to severe central sleep apnea and referred for implant of the remedē system / implanted with remedē system

Implant Exclusion Criteria:

* Patients meeting the criteria as referred to in the latest version of the implant manual

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with central sleep apnea
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stellbrink, Principal Investigator — Bielefeld-Klinikum; Stefan Anker, Principal Investigator — Herzzentrum Göttingen
Locations (10):
- Germany (7):
  - Herz- und Diabeteszentrum Bad Oeynhausen, Bad Oeynhausen
  - Klinikum Bielefeld Mitte, Bielefeld
  - Alice Hospital, Darmstadt
  - Albertinen Krankenhaus, Hamburg
  - Universitaetsklinikum Schleswig Holstein, Kiel
  - Klinikum Lünen - St Marien Hospital, Lünen
  - St. Vincenz-Krankenhaus, Paderborn
- Spain (3):
  - Hospital Infanta Cristina, Badajoz
  - Hospital Universitario de Burgos, Burgos
  - Hospital de Monteprincipe, Madrid

RESULTS

PARTICIPANT FLOW:
Groups:
- CSA Patients NOT Implanted With remedē System: For all patients diagnosed with CSA who will not move forward with remedē® system therapy, the intention is to obtain information on their alternate therapy, if any, and safety information, including all cause mortality and all cause hospitalizations during phone calls at 6, 12 and 24 months after enrollment.
Period: Overall Study
Arm/Group | CSA Patients NOT Implanted With remedē System | CSA Patients With remedē System
Started | 14 | 17
Completed | 0 (study terminated prematurely) | 0 (study terminated prematurely)
Not Completed | 14 | 17

BASELINE CHARACTERISTICS:
Groups:
- CSA Patients NOT Implanted With remedē® System: For all patients diagnosed with CSA who will not move forward with remedē® system therapy, the intention is to obtain information on their alternate therapy, if any, and safety information, including all cause mortality and all cause hospitalizations during phone calls at 6, 12 and 24 months after enrollment.
- CSA Patients With remedē System: For all patients diagnosed with CSA and referred for implant / or have already been implanted with remedē system, information from the implant procedure will be collected.
- Total: Total of all reporting groups
Arm/Group | CSA Patients NOT Implanted With remedē® System | CSA Patients With remedē System | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (6.8) | 69.2 (11.5) | 70.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  Germany | 12 | 16 | 28
  Spain | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of All Cause Mortality, SAEs, Stimulation Complaints, Device and/or Cardiovascular Related Events From Implant up to 5 Years.
Description: Collect short and long term clinical data on safety of the remede system implanted in daily practice.
  This outcome measure was intended to be collected up to 5 years, but at time of early study termination the data were only monitored until 24 months for 1 patient.
Time Frame: From implant up to 5 years (collected until 24 month FU)
Population: Viewing the limited amount of data at early study termination, the data should be interpreted with caution.
Measure: Count of Participants; unit: Participants
Arm/Group | CSA Patients With remedē System
Number analyzed (Participants) | 17
Participants
  Serious Adverse Events | 6
  Deaths | 0
  Serious Adverse Device Effects | 3
  Stimulation complaints | 1
  Cardiovascular events | 6

2. Secondary Outcome: Change in Apnea-hypopnea Index as Assessed by Polygraphy Compared to Baseline
Description: Evaluate changes in sleep study results at 12 months compared to baseline
Time Frame: 12 months post-implant
Population: A complete dataset is only available for 1 patient and due to confidentiality reasons for this 1 patient we prefer not to present this data.
Arm/Group | CSA Patients With remedē System
Number analyzed (Participants) | 0

3. Secondary Outcome: Impact on Quality of Life Compared to Baseline
Description: Evaluate impact on Quality of Life by using a general questionnaire, a sleep-specific questionnaire and a questionnaire specific for heart failure patients
Time Frame: Up to 5 years post-implant
Population: No data available on Quality of Life questionnaires; no patient completed the questionnaires at baseline AND at the 12M/24M follow-up at the time of premature study stop.
Arm/Group | CSA Patients With remedē System
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Reverse Remodelling Response as Assessed by Echo Compared to Baseline
Description: Evaluate reverse remodeling response in patients with reduced ejection fraction at baseline
Time Frame: 12 months post implant
Population: No data available; no patient had completed a 12 months echo prior to the premature study stop
Arm/Group | CSA Patients With remedē System
Number analyzed (Participants) | 0

5. Secondary Outcome: Incidence of All Cause Mortality and Hospitalizations up to 2 Years After Diagnosis of Central Sleep Apnea
Description: Collect site reported safety data on all patients diagnosed with central sleep apnea and not treated with the remede system
Time Frame: Up to 2 years (collected until 6M FU)
Population: No conclusion can be drawn on all-cause mortality and all-cause hospitalization rates for this group of patients;only 3 subjects diagnosed with CSA (not implanted) reached the 6M FU at the time of study termination. No deaths and/or hospitalizations had been reported in this subject group at the time of study termination.No 12M data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | CSA Patients NOT Implanted With remedē® System
Number analyzed (Participants) | 14
Participants
  hospitalizations | 0
  all cause mortality | 0

6. Other Pre Specified Outcome: Collect Clinical Characteristics and Symptoms of Patients With Central Sleep Apnea
Description: Characterstics and symptoms of patients screened for sleep disordered breathing were not collected and analyzed.
Time Frame: screening
Arm/Group | CSA Patients NOT Implanted With remedē® System | CSA Patients With remedē System
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | CSA Patients NOT Implanted With remedē® System | CSA Patients With remedē System
Serious Adverse Events (participants affected / at risk) | 0/14 | 6/17
Other Adverse Events (participants affected / at risk) | 0/14 | 4/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSA Patients NOT Implanted With remedē® System (N=14) | CSA Patients With remedē System (N=17)
Acute Reneal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) — One subject suffered from postoperative acute renal failure due to contrast fluid exposition at implant procedure
Cardiac Decompensation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac/cardiorespiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Other cardiac disorders (Cardiac disorders) | 0 (0) | 3 (4)
Lead Dislocation (Product Issues) | 0 (0) | 3 (3) — lead dislocations led to a system modification which was successful in all three patients, with one patient needing two modifications to achieve stable lead position
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSA Patients NOT Implanted With remedē® System (N=14) | CSA Patients With remedē System (N=17)
Diaphragm stimulation discomfort (General disorders) | 0 (0) | 1 (1)
Cardiac decompensation (Cardiac disorders) | 0 (0) | 1 (1)
beginning liver insufficiency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lead Dislocation (Product Issues) | 0 (0) | 1 (1) — 1 lead dislocation was not reported as SAE by site
atrial arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the early study termination, the amount of collected data was inconclusive at the time of early study termination to draw any conclusion on the study objectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The legal manufacturer of the medical device, Respicardia, shall be the owner of the Clinical study data including any results, and Respicardia shall have the right to control the publication timing, content and method for any public disclosure of the clinical study data. Respicardia's prior written approval must be obtained prior to any publication or disclosure of Clinical study data or results by Sponsor or Institution.